CLINICAL TRIAL: NCT05544630
Title: Effect of Aging on Postural Stability
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Zainab Ahmed Mahmoud, Resident Doctor at Audio vestibular Medicine Unit ENT Department, Al-Azhar University (Assiut), Sohag University
Other Study IDs: Soh-Med-22-07-16
Record Dates: First submitted 2022-09-13; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Effect of Aging on Postural Stability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: computerized dynamic posturography (sensory orgnization test) — assess of an individual's ability to maintain static and dynamic stance. The assessment is composed of a battery of tests that are similar to everyday conditions of daily living. There are four main components to CDP that are used clinically: the Sensory Organization Test (SOT),

SUMMARY:
Postural control of human body is a complex process involving visual , vestibular, somatosensory system and their central processing , add the vestibular system through its multiple connection coordinates movements of the head with movement of the eyes (to maintain clear vision ), trunk , and limbs (to maintain cephalic and postural stability ) via vestibulo-ocular and vestibulo-spinal reflexes respectively Global postural control shows alterations with aging increasing the chance of falls in the population aged 60 years or older, In older adults, poor postural balance can indicate an impaired ability to recover from small postural perturbations and be predictive of future falls

ELIGIBILITY:
Inclusion Criteria:

* Age: from 60 years to 80 years old.
* Sex: males and females
* All subject had no audio vestibular disease's.
* No evidence of cognitive dysfunction.
* No evidence of musculo-skeletal abnormalities.
* No motion intolerance.
* No history of any disease required to give treatment that could affect results

Exclusion Criteria:

* Old age person with cognitive dysfunction.
* Old age person with musculo-skeletal disorder.
* Adult person below age 60 years old.
* Old age person with neurological disease, motion intolerance, visual disorder, diabetes mellitus and hypertension.

Ages: 60 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: healthy ageing people not complaining imbalance not diabetic or hypertensive
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of change in balance function | 12 months
  Using computerized dynamic posturography ( sensory organization test)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baudry S. Aging Changes the Contribution of Spinal and Corticospinal Pathways to Control Balance. Exerc Sport Sci Rev. 2016 Jul;44(3):104-9. doi: 10.1249/JES.0000000000000080. No abstract available. PMID 27111478
- [Background] Haas BM, Burden AM. Validity of weight distribution and sway measurements of the Balance Performance Monitor. Physiother Res Int. 2000;5(1):19-32. doi: 10.1002/pri.181. PMID 10785908
- [Background] Henry M, Baudry S. Age-related changes in leg proprioception: implications for postural control. J Neurophysiol. 2019 Aug 1;122(2):525-538. doi: 10.1152/jn.00067.2019. Epub 2019 Jun 5. PMID 31166819
- [Background] Hu M, Chen T, Dong H, Wang W, Xu K, Lin P. [Clinical values of the sensory organization test in vestibular diseases]. Zhonghua Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2015 Sep;50(9):712-7. Chinese. PMID 26696341